CLINICAL TRIAL: NCT03199105
Title: Preoperative Education With Image Illustrations Enhances the Effect of Tetracaine Mucilage in Alleviating Postoperative Catheter-related Bladder Discomfort: a Prospective, Randomized, Controlled Study
Brief Title: Preoperative Education With Image Illustrations Enhances Effect of Tetracaine Mucilage in Alleviating Postoperative CRBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-159
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-06

CONDITIONS: Catheter Site Discomfort

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative education and tetracaine (Experimental)
  Interventions: Other: Preoperative education with image illustrations and/or local tetracaine mucilage
- tetracaine (Experimental)
  Interventions: Other: Preoperative education with image illustrations and/or local tetracaine mucilage

INTERVENTIONS:
Other: Preoperative education with image illustrations and/or local tetracaine mucilage — The patients were given preoperative education with image illustrations and/or local tetracaine mucilage to alleviate CRBD during the post-operative period.

SUMMARY:
Catheter-related bladder discomfort (CRBD) is not uncommon in male patients under general anesthesia, and it may cause patient agitation and exacerbated postoperative pain. In this study, the investigators will enroll male patients undergoing elective colonal and rectal surgery with surgical duration of at least 2 h, requiring catheterization of the urinary bladder with urinary catheterization after anesthetic induction, and compare preoperative education with image illustrations combined with local tetracaine mucilage vs. local tetracaine mucilage alone in alleviating CRBD during the post-operative period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years to 75 years.
2. American Society of Anesthesiologists (ASA) physical status I, II.
3. Undergoing elective noncardiac surgery with urinary catheterization after 4.anesthetic induction under general anesthesia.

5.Duration of surgery more than 2h 6.Glasgow Coma Scale (GCS) score of 15. Ability to communicate.

Exclusion Criteria:

1. History of bladder dysfunction, such as over active bladder (OAB, urinary frequency: more than three times in the night or more than eight times in 24 h).
2. History of bladder outflow obstruction.
3. Neurogenic bladder.
4. Impaired renal function.
5. Coagulopathy.
6. Known allergies to any anesthetic agent.
7. Family history of malignant hyperthermia.
8. Impairment of communication or cognition.
9. Psychopathy.
10. Active participation in another trial where the primary endpoint follow-up is ongoing.
11. Unwillingness or inability to comply with protocol procedures.

    -

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-10-20 (Estimated); Study Completion 2018-10-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative CRBD | 6 hours
  The incidence of postoperative CRBD; CRBD was assessed according to the following scaling system: no CRBD; mild CRBD (complaint about CRBD on questioning only); moderate CRBD (complaint about CRBD without enquiring); and severe CRBD (complaint about CRBD without enquiring, with urinary urgency demonstrated by a spontaneous behavioural response such as flailing limb, verbal responses, or attempt to remove the catheter)

SECONDARY OUTCOMES:
The severity of postoperative CRBD | 6 hours
  The severity of CRBD was assessed according to the following scaling system: no CRBD; mild CRBD (complaint about CRBD on questioning only); moderate CRBD (complaint about CRBD without enquiring); and severe CRBD (complaint about CRBD without enquiring, with urinary urgency demonstrated by a spontaneous behavioural response such as flailing limb, verbal responses, or attempt to remove the catheter)
The incidence of emergence agitation | 6 hours
  Using Riker Sedation-Agitation Scale, where 5 to 7 represents agitation and 1 to 3 represents deep sedation
The incidence of postoperative pain | 6 hours
  The incidence of postoperative pain;Using a visual analog scale (VAS) score of 0-10, where 0 represents no pain and 10 represents worst imaginable pain.
The severity of postoperative pain | 6 hours
  Using a visual analog scale (VAS) score of 0-10, where 0 represents no pain and 10 represents worst imaginable pain.
Incidenc of adverse events | 6 hours
  Incidenc of adverse events, such asrespiratory depression (SpO2<90%), deep sedation, and toxicity of tetracaine

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Zhou L, Zhou L, Tian L, Zhu D, Chen Z, Zheng C, Zhou T, Zeng X, Jiang X, Jiang C, Bo L. Preoperative education with image illustrations enhances the effect of tetracaine mucilage in alleviating postoperative catheter-related bladder discomfort: a prospective, randomized, controlled study. BMC Anesthesiol. 2018 Dec 22;18(1):204. doi: 10.1186/s12871-018-0653-y. PMID 30579342